CLINICAL TRIAL: NCT03871361
Title: Abatacept in Patients With Birdshot HLA A29 Uveitis: A Phase II Prospective 0pen Label Interventional Proof-of-Concept Study
Brief Title: Abatacept in Patients With Birdshot HLA A29 Uveitis
Acronym: HLA-A29
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Ziekenhuis Netwerk Antwerpen (ZNA) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S62092; 2018-003653-16 (EudraCT Number); IM101-794 (Other Grant/Funding Number: BMS)
Record Dates: First submitted 2019-03-05; First posted 2019-03-12 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Eye Diseases; Uveitis
Keywords: Birdshot Uveitis; HLA A29; Abatacept
MeSH Terms: conditions — Eye Diseases; Uveitis | interventions — Abatacept

STUDY DESIGN:
Intervention Model Description: Prospective 0pen Label Interventional Proof-of-Concept Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Abatacept 125 MG/ML Prefilled Syringe (Experimental): Participants will inject the drug at home on a weekly basis. Participants will receive the syringes on the visit dates, supplying them for the period until the next visit. At baseline, participants will be explained and shown how to inject the drug themselves.
  Subject will have to stop all concomitant immunosuppressive drugs at baseline, e.g. Corticosteroids, Methotrexate, Mofetil Mycophenolate, Azathioprine, Tacrolimus, Sirolimus or Cyclosporin. Other drugs can be continued. In case of recurrence in the abatacept group, the study will end for that subject.
  Patients treated with abatacept (ORENCIA) may receive concurrent vaccinations, except for live vaccines. Live vaccines should not be given concurrently with abatacept or within 3 months of its discontinuation.
  Interventions: Drug: Abatacept 125 MG/ML Prefilled Syringe

INTERVENTIONS:
Drug: Abatacept 125 MG/ML Prefilled Syringe — Abatacept 125 MG/ML Prefilled Syringe [Orencia] weekly
  Other Names: Orencia

SUMMARY:
To assess the efficacy and safety of Abatacept as an immunosuppressive treatment in Birdshot uveitis. The primary objective is to test the efficacy to suppress inflammation in active Birdshot uveitis patients, using quantitative and qualitative measurements of visual function.

DETAILED DESCRIPTION:
To assess the efficacy and safety of Abatacept as an immunosuppressive treatment in Birdshot uveitis. The primary objective is to assess the efficacy to suppress active uveitis in Birdshot uveitis and to induce inflammatory remission during the 1 year treatment and after 2 years of treatment. Treatment efficacy will be assessed, using quantitative and qualitative measurements of visual function. In this trial we will also assess the utility of quantitative outcome measures in detecting disease activity.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age.
2. Subject is diagnosed with Birdshot uveitis, HLA A 29+
3. Subject must have active disease at the Baseline visit as defined by the presence of at least 1 of the following parameters in at least one eye :

   -Active, inflammatory, chorioretinal and/or inflammatory retinal vascular lesions

   -≥ 1+ vitreous haze (National Eye Institute [NEI]/SUN criteria)
4. Subjects who do not have previous, active or latent tuberculosis (TB). Subjects with negative QuantiFERON®-TB Gold test (or interferon-gamma release assay (IGRA) equivalent) are eligible. Subjects with a repeat indeterminate QuantiFERON®-TB Gold test (or IGRA equivalent) result are not eligible. The TB screening tests are diagnostic tests. In the event of a negative TB screening test, the results are to be interpreted in the context of the patient's epidemiology, history, exam findings, etc. and it is the responsibility of the investigator to determine if a patient has previous, active or latent tuberculosis or not. Under no circumstances can a patient with a positive QuantiFERON®-TB Gold test (or IGRA equivalent) enter the study.

Exclusion Criteria:

1. Subject with prior inadequate response to high-dose oral corticosteroids (>30 mg of prednisolone or equivalent)
2. Subject with confirmed or suspected infectious uveitis, including but not limited to infectious uveitis due to TB, cytomegalovirus (CMV), Human T-Lymphotropic Virus Type 1 (HTLV-1), Whipple's disease, Herpes Zoster virus (HZV), Lyme disease, toxoplasmosis and herpes simplex virus (HSV).
3. Subject with corneal or lens opacity that precludes visualization of the fundus or that likely requires cataract surgery during the duration of the trial.
4. Subject with intraocular pressure of ≥ 25 mmHg and on ≥ 2 glaucoma medications or evidence of glaucomatous optic nerve injury.
5. Subject with Best Corrected Visual Acuity (BCVA) less than 20 letters (Early Treatment Diabetic Retinopathy Study) in at least one eye at the Baseline Visit.
6. Subject with intermediate uveitis or panuveitis that has signs of intermediate uveitis (e.g.presence or history of snowbanking or snowballs) and symptoms and/or magnetic resonance imaging (MRI) findings suggestive of a demyelinating disease such as multiple sclerosis. All subjects with intermediate uveitis or panuveitis that have signs of intermediate uveitis (e.g., presence or history of snowbanking or snowballs) must have had a brain MRI within 90 days prior to the Baseline Visit.
7. Subject has had previous exposure to anti-tumor necrosis factor (TNF) therapy or any biologic therapy (except intravitreal anti-vascular endothelial growth factor [VEGF] therapy) with a potential therapeutic impact on non-infectious uveitis
8. Subject with exposure to classic immunosuppressive therapy, in which the dose has been increased within the last 28 days prior to Baseline visit or is within the following doses at the screening visit: Methotrexate (MTX) >25 mg per week Cyclosporine > 4 mg/kg per day Mycophenolate mofetil >2 grams per day or an equivalent drug to mycophenolate mofetil (e.g. mycophenolic acid) at an equivalent dose approved by the Medical Monitor. Azathioprine > 175 mg per day Tacrolimus (oral formulation) >8 mg per day.
9. Subject is still on immunosuppressive therapy ( Corticosteroids, Methotrexate, Cyclosporine, Mycophenolate Mofetil, Azathioprine, Tacrolimus, Sirolimus) at the baseline visit.
10. Subject has received Iluvien® (glucocorticosteroids implant) within 3 years prior to the Baseline visit or that has had complications related to the device. Subject has had Iluvien® (glucocorticosteroids implant) removed within 90 days prior to the Baseline visit or has had complications related to the removal of the device.
11. Subject has received intraocular or periocular corticosteroids within 30 days prior to Baseline visit.
12. Subject with proliferative or severe non-proliferative diabetic retinopathy or clinically significant macular edema due to diabetic retinopathy. Subject with neovascular/wet age-related macular degeneration Subject with abnormality of vitreo-retinal interface (i.e., vitreomacular traction, epiretinal membranes, etc.) with the potential for macular structural damage independent of the inflammatory process. Subject with severe vitreous haze that precludes visualization of the fundus at the Baseline visit.
13. Subject has received Ozurdex® (dexamethasone implant) within 6 months prior to the Baseline visit. Subject has received intravitreal anti-VEGF therapy within 45 days of the Baseline visit for Lucentis® (ranibizumab) or Avastin® (bevacizumab) or within 60 days of the Baseline visit for anti-VEGF Trap (aflibercept).
14. Subject has received intravitreal methotrexate within 90 days prior to the Baseline visit
15. Subject on systemic carbonic anhydrase inhibitor within 1 week prior to Screening visit.
16. Subject with macular edema as the only sign of uveitis.
17. Subject with a history of scleritis.
18. Subject on cyclophosphamide within 30 days prior to the Baseline visit.
19. Subjects with a known HIV, HepB/C infection.
20. Subjects with an active or recent acute infection.
21. Subjects with a history of chronic or recurrent bacterial, viral or systemic fungal infections.
22. Subjects with malignancies.
23. Subjects who have received any live vaccines within 3 months of the start of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
time to recurrence in ≥1 eye | 1 year and 2 years
  Patients are assessed for recurrence, if at least 1 of the following criteria are fulfilled in at least 1 eye.
  * worsening of BCVA (Best Corrected Visual Acuity measured by ETDRS chart) by >15 letters relative to baseline
  * 30% increase of central retinal thickness on OCT (Optical Coherence Tomography) relative to baseline
  * 2-step increase in VH (Vitreous Haze) grade relative to baseline
  * new active, inflammatory choroidal (detected on ICG Angiography) and/or inflammatory retinal vascular lesions relative to baseline (detected on FA: fluorescein angiography).

SECONDARY OUTCOMES:
Change in Vitreous Haze (VH) Grade in Each Eye From Baseline to the Final/Early Termination Visit | 1 year and 2 years
  Vitreous haze is measured using dilated indirect ophthalmoscopy (DIO) and assessed by the Investigator according to National Eye Institute (NEI) and SUN criteria:
  Grade 0: No evident vitreous haze Grade 0.5+: Slight blurring of the optic disc margin because of the haze; normal striations and reflex of the nerve fiber layer cannot be visualized; Grade 1+: Permits a better definition of both the optic nerve head and the retinal vessels (compared to higher grades); Grade 2+: Permits better visualization of the retinal vessels (compared to higher grades); Grade 3+: Permits the observer to see the optic nerve head, but the borders are quite blurry; Grade 4+: Optic nerve head is obscured.
Change In Logarithm of the Minimum Angle of Resolution (LogMAR) Best Corrected Visual Acuity (BCVA) In Each Eye From Baseline to the Final/Early Termination Visit | 1 year and 2 years
  Using corrective lenses based on that visit's refraction testing, participant's best corrected visual acuity is measured using an Early Treatment Diabetic Retinopathy Study (ETDRS) logMAR chart.
Time to Optical Coherence Tomography (OCT) Evidence of Macular Edema in At Least 1 Eye On or After Baseline | 1 year and 2 years
  Optical coherence tomography is performed at every visit using the Zeiss Cirrus OCT. Images are evaluated by a central reader (PI). Macular edema is defined as cystoid macular edema. OCT evidence of macular edema on or after Baseline is to be counted as an event. Dropouts due to reasons other than OCT evidence of macular edema are to be considered as censored observations at the time of dropping out.
  Optical Coherence Tomography will be measured using the Zeiss Cirrus OCT. For each eye a macular cube slab 512x128 and 2 HD 5 lines rasters (1 on 180° and 1 on 90°) will be taken, centered on the fovea.
Percent Change in Central Retinal Thickness in Each Eye From Baseline to the Final/Early Termination Visit | 1 year and 2 years
  Optical coherence tomography is performed at every visit using the Zeiss Cirrus OCT.Retinal thickness will be measured on the macular cube slab centered on the fovea. This will be measured by a central reader (PI).
Percent Change in Choroidal Thickness in Each Eye From Best State Achieved Prior to week 6 to the Final/Early Termination Visit | 1 year and 2 years
  Choroidal thickness will be measured using the EDI mode of the Zeiss Cirrus OCT (HD 5 lines raster) and will be measured by a central reader (PI).
Change in Visual Functioning Questionnaire 25 (VFQ-25) Composite Score From Baseline to the Final/Early Termination Visit | 1 year and 2 years
  The National Eye Institute VFQ-25 is an ocular disease-specific survey that measures the influence of visual disability and visual symptoms on generic health domains such as emotional well-being and social functioning, in addition to task-oriented domains related to daily visual functioning
Change in scoring of Dual Fluorescein and ICG (Indocyanine Green) angiography from best state achieved | 1 year and 2 years
  Change in scoring of Dual Fluorescein and ICG (Indocyanine Green) angiography from best state achieved, as defined by the Angiography Scoring for Uveitis Working group using the Heidelberg Scanning LASER fluorescein and ICG angiography
Change in Full Field ElectroRetinoGraphy (ERG) using the ISCEV standard protocols from baseline until the Final Visit | 1 year and 2 years
  Quantitative values, such as 30 Hz implicit time, amplitude in a and b wave and latency will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Pieter-Paul FA Schauwvlieghe, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZLeuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schauwvlieghe PP, Van Calster J, Herbort CP Jr, Kestelyn PA, de Vlam K. Efficacy and safety of abatacept to treat active birdshot uveitis: a prospective open label interventional proof-of-concept trial. Br J Ophthalmol. 2024 Jan 29;108(2):244-252. doi: 10.1136/bjo-2022-321585. PMID 36585127
- See also: Belgian Dataprotection Authority — http://www.gegevensbeschermingsautoriteit.be